CLINICAL TRIAL: NCT02203396
Title: A Single-Arm Phase 2 Study With Optimized Standard Protocol for Severe Aplastic Anemia
Acronym: OSP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2014006
Record Dates: First submitted 2014-07-27; First posted 2014-07-29 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2024-05

CONDITIONS: Aplastic Anemia
Keywords: SAA; Immunosuppressive treatment; ATG; Cyclosporine; Levamisole
MeSH Terms: conditions — Anemia, Aplastic | interventions — thymoglobulin; Cyclosporine; Levamisole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Severe Aplastic Anemia (Experimental): Drug: rabbit ATG, Cyclosporine, Levamisole
  Interventions: Drug: rabbit ATG, Cyclosporine, Levamisole

INTERVENTIONS:
Drug: rabbit ATG, Cyclosporine, Levamisole — rATG is administered at a dose of 1.97 mg/kg/day for 9 days CSA is administered orally at a dose of 3 mg/kg qod Levamisole is administered orally at a dose of 2.5 mg/kg qod. The CSA and LMS is designed to alternately every other day.
  Other Names: rATG; CSA; LMS

SUMMARY:
Severe acquired aplastic anaemia (SAA) is a bone marrow failure disease characterized by pancytopenia and a hypocellular bone marrow. The corn pathophysiological mechanism is the destruction of hematopoietic stem/progenitor cells mediated by auto-reactive effector T cells. Immunosuppressive therapy with horse antithymocyte globulin (ATG) plus cyclosporine (CSA) is currently the standard of treatment in patients with aplastic anaemia who are not eligible for bone marrow transplantation and with response rates from 40% to 70%. Previous studies showed that horse ATG (hATG) is apparently more effective than rabbit ATG (rATG) as the latter has higher treatment related mortality (TRM). Unfortunately hATG is unavailable in China, so we conduct a optimized standard treatment (9 days protocol) of rATG plus CSA and Levamisole (LMS) Sequential maintaining (termed Optimized Standard Protocol, OSP) for severe aplastic anemia. This prospective study is designed to evaluate the efficacy and safety of Optimized Standard Protocol as first line therapy in newly diagnosed severe aplastic anemia patients.

DETAILED DESCRIPTION:
During the treatment period, rATG is administered at a dose of 1.97 mg/kg/day for 9 days by slow intravenous infusion. CSA is administered orally at a dose of 3 mg/kg qod, and Levamisole was administered orally at a dose of 2.5 mg/kg qod. The CSA and Levamisole (LMS) is designed to alternately every other day.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed SAA (according to the standard criteria)

  1. Bone marrow cellularity less than 30% (excluding lymphocytes)
  2. At least two of the following: Absolute neutrophil count less than 500/ uL; Platelet count less than 20,000/ uL; Absolute reticulocyte count less than 20,000/ uL.
* Age greater than or equal to 6 years old

Exclusion Criteria:

* Serum creatinine greater than 2.5 mg/dL
* Underlying carcinoma (except local cervical, basal cell, squamous cell)
* Prior immunosuppressive therapy with ATG, antilymphocyte globulin (ALG), or high dose cyclophosphamide.
* Current pregnancy or lactation or unwillingness to take oral contraceptives or use an effective method of birth control.
* Diagnosis of Fanconi anemia or other congenital bone marrow failure syndromes
* Evidence of a clonal disorder on cytogenetics. Patients with super severe neutropenia (ANC less than 200/uL) will not be excluded if results of cytogenetics are not available or pending.
* Underlying immunodeficiency state including seropositivity for HIV
* Inability to understand the investigational nature of the study or give informed consent
* Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy, or that death within 7-10 days is likely.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
the response and complete remission rate with Optimized Standard Protocol. | month +6
  Response will be evaluated at each clinic visit. Complete response (CR) was defined as achieving all three peripheral blood count criteria: (1) Hb level up to the normal range; (2) ANC≥1.5×109/L; (3) PLT≥100×109/L.
  Partial response (PR) was defined as transfusion independent, no longer meeting criteria for severe disease. Persistence of transfusion requirement or death was evidence of no response (NR).

SECONDARY OUTCOMES:
Relapse rate, sustained response (SR), survival, and clonal evolution to myelodysplasia and acute leukemia. | month +12, month +60
  Relapse was defined as a responder who met criteria for SAA again after achieving response and keeping stable blood counts for at least 3 months.
  Sustained response (SR) was defined as Hb > 10 g/dL at month +12 and +60, in the absence of any treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Yizhou, M.D., Ph.D, Principal Investigator — Anemia Therapeutic Center, Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Result] Rosenfeld S, Follmann D, Nunez O, Young NS. Antithymocyte globulin and cyclosporine for severe aplastic anemia: association between hematologic response and long-term outcome. JAMA. 2003 Mar 5;289(9):1130-5. doi: 10.1001/jama.289.9.1130. PMID 12622583
- [Result] Camitta BM, Rappeport JM, Parkman R, Nathan DG. Selection of patients for bone marrow transplantation in severe aplastic anemia. Blood. 1975 Mar;45(3):355-63. PMID 1090310